CLINICAL TRIAL: NCT05821569
Title: Cerebral Synchronization Between Mothers and Their Newborns During Breastfeeding and Related Oxytocin Response, According to Different Reciprocal Positioning of the Dyad, and Possible Related Benefit for Postpartum Depressive Symptoms
Brief Title: Cerebral Synchronization Between Mothers and Their Newborns During Breastfeeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 53/22
Record Dates: First submitted 2023-03-24; First posted 2023-04-20 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Depression, Postpartum
Keywords: Breastfeeding; Near-infrared spectroscopy; Postpartum depression
MeSH Terms: conditions — Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard position during breastfeeding: Women who adopted, according to their preference and/or to the professional advice and support of the nursing staff the standard position (derived from UNICEF guidelines) to breastfeed
  Interventions: Other: Standard approach
- biological nurturing: Women who adopted, according to their preference and/or to the professional advice and support of the nursing staff, the biological nurturing approach to breastfeed
  Interventions: Other: Biological nurturing

INTERVENTIONS:
Other: Standard approach — Adoption of standard approach (derived by Unicef guidelines) to breastfeed
  Groups: standard position during breastfeeding
Other: Biological nurturing — Adoption of biological nurturing approach to breastfeed
  Groups: biological nurturing

SUMMARY:
Different reciprocal positions of mother and newborn during breastfeeding may be adopted. Other than the one derived from UNICEF guidelines, or standard position, an approach called biological nurturing has been recently proposed. It aims to promote the activation of neonatal primitive reflexes, breast problems reduction (e.g. cracked or sore nipple) and, overall, spontaneity and naturalness of mother-newborn dyad behaviour during feeding.

The study of newborn cortical activation by functional near-infrared spectroscopy (fNIRS), a safe and minimally invasive functional neuroimaging technique based on haemoglobin absorption of near-infrared light, showed that baby's cortex exhibit a wide activation associated with breastfeeding. Moreover, preliminary and not yet published data, collected by fNIRS hyperscanning (e.g. the simultaneous detection of brain functional activation from two individuals living the same experience) in the Nursery of our Institute, evidenced that mother-newborn dyads adopting a biological nurturing approach to breastfeeding show a neural synchronization between their frontal cortex during such experience. Basing on this new evidence, it is now worth to understand if a biological nurturing approach to breastfeeding may promote such neural synchronization, even when postpartum depressive symptoms are present. Accordingly, biological nurturing may result to be protective for the neural basis of mother-newborn relationship, also in case of a postnatal affective suffering and helping to prevent its potential long term consequences on maternal wellbeing and infant neurodevelopment as well. Moreover, since oxytocin is a neuropeptide with widespread influence on parental function, including lactation and nurturing maternal behaviour physiology, if a biological nurturing approach to breastfeeding may promote the oxytocin level in the mother and/or in the newborn is worth to understand as well, taking into account again possible relations with postpartum depression symptoms. the aim of this study is to evaluate, by fNIRS hyperscanning, if the frontal cerebral cortex functional synchronization of mother-newborn dyads, who adopt a reciprocal positioning according to the biological nurturing approach during breastfeeding, differs from that of mother-newborn dyads adopting the standard position, taking into account the intensity of mother's postpartum depressive symptoms.

DETAILED DESCRIPTION:
Breastfeeding is a very important experience since the beginning of life, supplying the best physical, biological and affective conditions for newborn's growth and development. Its promotion of motor, cognitive (e.g. language, memory), and emotional development in the long term was also observed. Benefits are for the mother too, including a reduction of the risk for postpartum depression. This clinical condition is the most common maternal psychiatric disorder after childbirth, observed in 10%-15% of mothers, and may adversely affect mother-newborn relationship, psychophysical maternal wellbeing, and infant development.

Different reciprocal positions of mother and newborn during breastfeeding may be adopted. Other than the one derived from UNICEF guidelines, or standard position, an approach called biological nurturing has been recently proposed. It aims to promote the activation of neonatal primitive reflexes, breast problems reduction (e.g. cracked or sore nipple) and, overall, spontaneity and naturalness of mother-newborn dyad behaviour during feeding.

Newborn cortical activation associated with breastfeeding was studied too. By functional near-infrared spectroscopy (fNIRS), a safe and minimally invasive functional neuroimaging technique based on haemoglobin absorption of near-infrared light, our research group showed that baby's cortex exhibit a wide activation associated with breastfeeding. Moreover, preliminary and not yet published data, collected by fNIRS hyperscanning (e.g. the simultaneous detection of brain functional activation from two individuals living the same experience) in the Nursery of our Institute, evidenced that mother-newborn dyads adopting a biological nurturing approach to breastfeeding show a neural synchronization between their frontal cortex during such experience. Basing on this new evidence, it is now worth to understand if a biological nurturing approach to breastfeeding may promote such neural synchronization, even when postpartum depressive symptoms are present. Accordingly, biological nurturing may result to be protective for the neural basis of mother-newborn relationship, also in case of a postnatal affective suffering and helping to prevent its potential long term consequences on maternal wellbeing and infant neurodevelopment as well. Moreover, since oxytocin is a neuropeptide with widespread influence on parental function, including lactation and nurturing maternal behaviour physiology, if a biological nurturing approach to breastfeeding may promote the oxytocin level in the mother and/or in the newborn is worth to understand as well, taking into account again possible relations with postpartum depression symptoms. the aim of this study is to evaluate, by fNIRS hyperscanning, if the frontal cerebral cortex functional synchronization of mother-newborn dyads, who adopt a reciprocal positioning according to the biological nurturing approach during breastfeeding, differs from that of mother-newborn dyads adopting the standard position, taking into account the intensity of mother's postpartum depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Full term healthy newborn
2. Weight > 2500 gr
3. Vaginal delivery
4. Breastfeeding already started
5. Absence of breast problems (e.g. cracked or sore nipple)
6. Parents' consent to research participation

Exclusion Criteria:

1. Syndromic diagnosis (genetic/hereditary)
2. Condition affecting a major organ (heart disease, cerebropathy, etc.)
3. Medication intake that may interfere with the data collection (e.g. analgesics)
4. Newborn head lesion that may interfere with the fNIRS assessment (e.g. due to an operative delivery)
5. Mother history of neurological or neurosensory disorder, psychosis, bipolar disorder, and substance abuse or addiction.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Full term healthy newborns and their mothers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
To compare the frontal cerebral cortex functional synchronization in mother-newborn dyads adopting biological nurturing vs standard position to breastfeed | At the second day after birth
  To evaluate by fNIRS hyperscanning if the frontal cerebral cortex functional synchronization of mother-newborn dyads who adopt a reciprocal positioning according to the biological nurturing approach during breastfeeding, differs from that of mother-newborn dyads adopting the standard position. Cortical activation associated with breastfeeding will be assessed by multichannel fNIRS (Hitachi mod. ETG 4000, 48 channels), using a fibre holder in plastic in mothers and in soft material (neoprene) in newborns, with an interfibre distance of 3 cm. Bilateral functional activity in the frontal and somatomotor areas will be monitored in both mother and newborn (24 channels each).
To compare the presence of postpartum depressive symptoms in women adopting biological nurturing vs standard position to breastfeed | At the second day after birth
  The presence of maternal postpartum depressive symptoms will be evaluated by the Edinburgh Postnatal Depression Scale (EPDS), a set of 10 screening questions. Each answer is given a score of 0 to 3. Cut-off values of 10 or higher suggest the presence of depression.

SECONDARY OUTCOMES:
To compare the oxytocin level of mothers adopting different position during breastfeeding (standard position vs biological nursing) | At the second day after birth
  To evaluate differences in salivary oxytocin levels of mothers adopting the biological nurturing approach to breastfeed vs mothers adopting the standard position. In multivariate analysis also the intensity of maternal postpartum depressive symptoms assessed by EPDS will be take into account. EPDS is a set of 10 screening questions. Each answer is given a score of 0 to 3. Cut-off values of 10 or higher suggest the presence of maternal postpartum depression.
To evaluate the oxytocin level of newborns according to different position adopted during breastfeeding (standard position vs biological nursing) | At the second day after birth
  To evaluate differences in salivary oxytocin levels of newborns breastfed adopting the biological nurturing approach vs newborns breastfed adopting the standard position

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bembich, MSC, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy